CLINICAL TRIAL: NCT04041232
Title: Evaluation of Glycerol Phenylbutyrate (PBA) Use in Endoplasmic Reticulum Stress Reduction in ATF6-/- Patients
Brief Title: PBA Use for Treatment of ATF6-/- Patients
Status: Suspended | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Administrative changes
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAR9833
Record Dates: First submitted 2019-07-31; First posted 2019-08-01 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: ACHROMATOPSIA 7; Achromatopsia
Keywords: achromatopsia; PBA; ATF6; color blindness
MeSH Terms: conditions — Color Vision Defects | interventions — glycerol phenylbutyrate

STUDY DESIGN:
Intervention Model Description: Two patients will receive PBA as treatment for ATF6-/- Achromatopsia.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- PBA treatment of ATF6-/- Achromatopsia (Experimental): Patients will be monitored at the baseline visit, followed by a second and third visit that will be 1 and 3 months after the initial visit. Patients will complete a standard visual functioning questionnaire and undergo a complete ophthalmic evaluation at each visit. Other visual assessments will consist of color vision testing, contrast sensitivity, retinal imaging, and macular sensitivity testing using microperimetry. Full-field electroretinogram will also be performed at the baseline visit and after 1 and 3 months of PBA use. If improvement in retinal function is observed, an additional ophthalmic evaluation will be conducted after 6 months of PBA use. A blood draw will be performed at each visit to test for any indications of adverse effects from drug use.
  Interventions: Drug: PBA

INTERVENTIONS:
Drug: PBA — Glycerol phenylbutyrate (PBA) is a triglyceride that consists of three molecules of phenylbutyrate linked to a glycerol backbone. It is a nitrogen-binding agent that has been approved by the Food and Drug Administration (FDA) for the treatment of urea cycle disorders. Oral supplementation of PBA demonstrated no severe side effects, and are found to be therapeutically effective in reducing ER stress. Patients will be instructed to take three doses of PBA per day at equally divided time intervals and rounded up to the nearest 0.5 mL. The total dose of PBA will be 4.5 to 11.2 mL/m2/day (5 to 12.4 g/m2/day) and will not exceed 17.5 mL/day (19 g/day).
  Other Names: Glycerol Phenylbutyrate

SUMMARY:
Some patients with achromatopsia, an inherited disorder characterized by partial or complete loss of color vision, carry mutations in ATF6. ATF6 is a gene that is responsible for coding a protein that acts in response to endoplasmic reticulum (ER) stress. When the ATF6 protein is mutated, retinal function decreases, contributing to color blindness. The study aims to investigate whether an already FDA-approved drug, glycerol phenylbutyrate (PBA), can improve retinal function inpatients with achromatopsia caused by ATF6 mutations. Patients will be instructed to take three doses of PBA per day at equally divided time intervals and rounded up to the nearest 0.5 mL. The total dose of PBA will be 4.5 to 11.2 mL/m2/day (5 to 12.4 g/m2/day) and will not exceed 17.5 mL/day (19 g/day). Their condition will be monitored over the course of a minimum of 3 clinic visits that will consist of a number of retinal function tests, fundus examinations, and imaging procedures. Findings from the study could elucidate the potential for PBA to serve as a treatment for patients with ATF6-mediated a chromatopsia.

DETAILED DESCRIPTION:
ATF6 has been described as an endoplasmic reticulum (ER) stress-regulated transmembrane protein that activates the transcription of molecular chaperones in response to ER stress. Patients harboring mutations in ATF6 present with decreased retinal function and are diagnosed with achromatopsia. The investigator's research group has previously demonstrated that administration of glycerol phenylbutyrate (PBA), a fatty acid compound that facilitates protein folding, can lead to enhanced retinal function in mice that are homozygous for the ATF6 mutation. This study will investigate the effects of PBA administration in two patients who carry ATF6-/- mutations and a diagnosis of achromatopsia. Enrolled subjects will undergo a minimum of 3 clinic visits that consist of a complete ophthalmic examination (best-corrected visual acuity, intraocular pressure, anterior segment examination, slit lamp and binocular fundus examination), a visual functioning questionnaire, color vision tests, contrast sensitivity tests, retinal imaging (optical coherence tomography, short wavelength autofluorescence and near-infrared autofluorescence), a macular sensitivity test (Nidek microperimetry) and full-field electroretinogram (ffERG). A blood draw will be performed at each visit to test for any indications of adverse effects from drug use. Subjects will be instructed to take 3 doses of PBA per day, totaling to a dose of 4.5 to 11.2 mL/m2/day (5 to 12.4 g/m2/day).

ELIGIBILITY:
Inclusion Criteria:

* Patients harboring mutations in ATF6 present with decreased retinal function

Exclusion Criteria:

* Patients who are minors
* Patients who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2025-04-08 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Changes in best corrected visual acuity (BCVA) | Baseline, 1 month, 3 months, 6 months post-PBA use
  to measure changes in vision at each time point
Changes in contrast sensitivity | Baseline, 1 month, 3 months, 6 months post-PBA use
  using Pelli Robson charts
Changes in color vision | Baseline, 1 month, 3 months, 6 months post-PBA use
  using D50
Changes in macular sensitivity | Baseline, 1 month, 3 months, 6 months post-PBA use
  using microperimetry (Nidek)
Changes in retinal imaging | After 1 and 3 months of PBA use. If changes in retinal function is observed, an additional ophthalmic evaluation will be conducted after 6 months of PBA use
  including optical coherence tomography (OCT), short wavelength autofluorescence (SW-AF), and near-infrared autofluorescence (NIR-AF)
Changes in Full-field Electroretinogram (ffERG) X | After 1 and 3 months of PBA use. If changes in retinal function is observed, an additional ophthalmic evaluation will be conducted after 6 months of PBA use
  to measure changes in rod and cone traces

SECONDARY OUTCOMES:
Changes in intraocular pressure | Baseline, 1 month, 3 months, 6 months post-PBA use
  part of full ophthalmic evaluation
Changes in anterior segment | After 1 and 3 months of PBA use. If changes in retinal function is observed, an additional ophthalmic evaluation will be conducted after 6 months of PBA use
  part of full ophthalmic evaluation
Changes observed in posterior segment (slit lamp and binocular fundus examination) | After 1 and 3 months of PBA use. If changes in retinal function is observed, an additional ophthalmic evaluation will be conducted after 6 months of PBA use
  part of full ophthalmic evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Tsang, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States